CLINICAL TRIAL: NCT02595827
Title: Universal Versus Conditional Follow Up for Children With Unclassified Fever at the Community Level: A Cluster-Randomized, Community-based, Non-Inferiority Trial in Kalemie, Democratic Republic of Congo (DRC)
Brief Title: Non-inferiority Trial of Conditional vs Universal Follow up for Children With Fever in Democratic Republic of Congo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: International Rescue Committee (Other); University Research Co, LLC (Industry); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 68295
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Fever
Keywords: Pediatrics; Epidemiology; Fever; Democratic Republic of the Congo; Randomized Controlled Trial
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Universal (No Intervention): In this group, caretakers of children will receive the standard advice under current iCCM guidelines in DRC. Specifically, the CHW will advise that the child come back in 2-3 days.
- Conditional (Active Comparator): In this Conditional Advice group, caretakers will be given advice that is modified from the current iCCM guidelines. Specifically, the CHW will advise that the child come back in 2-3 days if the child's symptoms continue.
  Interventions: Other: Conditional Advice

INTERVENTIONS:
Other: Conditional Advice — Caretakers are told to return in 2-3 only (Conditional Advice) if the child's symptoms continue.
  Arms: Conditional

SUMMARY:
Providers in integrated Community Case Management (iCCM) programs in low resource settings often see children without any danger signs, presenting with fever but not having pneumonia, malaria, or diarrhea. These children are sent home (often with analgesic only), and caretakers are advised to return in 2 or 3 days. In this study, we are evaluating if conditional return advice (i.e. return in 2 or 3 day only if your child is still sick") results in the same proportion of children remaining with fever one week after identification, as the current universal return advice.

DETAILED DESCRIPTION:
Fevers in childhood are common and usually self resolve. In rural Democratic Republic of Congo (and many other settings), when a febrile child presents to a community health worker (CHW), the child is assessed for malaria, pneumonia, and diarrhea, and other danger signs, according to World Health Organization (WHO) guidelines for integrated Community Case Management (iCCM) of childhood illnesses. In the cases where 1) there are no danger signs present, and 2) malaria, pneumonia, and diarrhea have been ruled out, the CHW provides an antipyretic only, sends the child home, and advises all such cases to come back in 3 days. We hypothesize, however, that health outcomes for these cases will be equivalent if the CHW advises to come back in 3 days, only if symptoms have not resolved.

To test this hypothesis, we are conducting a cluster-randomized, community-based non-inferiority trial in two zones of Kalemie, Katanga Province, Democratic Republic of Congo. In this area, the International Rescue Committee (IRC) has been supporting the training, scale-up, and rollout of community health workers who conduct iCCM as per WHO guidelines and with Ministry of Health oversight. CHWs have unique non-overlapping catchment areas, and groups of CHWs (average 5-7) are associated with health clinics. We will utilize this group structure as the unit of randomization; health clinics (and thereby, groups of CHWs) will be randomly allocated to one of two groups in terms of the advice given to caretakers of children who have no danger signs, have neither malaria, pneumonia, nor diarrhea, and are thus classified as having fever of non-identified origin.

* Group 1 (Universal follow-up): CHWs in this group will advise caretakers to follow up in 3 days
* Group 2 (Conditional follow-up): CHWs in this group will advise caretakers to follow up in 3 days if symptoms/signs remain the same (or worsen).

ELIGIBILITY:
Inclusion Criteria:

* Agree to recruitment script provided by CHWs at the time of identification of eligible

Exclusion Criteria:

* None

Ages: 2 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4451 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2016-12-05 (Actual)

PRIMARY OUTCOMES:
Clinical failure at 7 days | 1 week
  If the child has fever, has a CHW-treatable condition (pneumonia, malaria, or diarrhea), or is referred for care at the Day 7 visit, the child has met the definition of the primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Luke C Mullany, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- International Rescue Committee, Kalemie Office, Kalemie, Katanga, Democratic Republic of the Congo

REFERENCES:
- [Derived] Mullany LC, van Boetzelaer EW, Gutman JR, Steinhardt LC, Ngoy P, Barbera Lainez Y, Wittcoff A, Harvey SA, Ho LS. Universal versus conditional day 3 follow-up for children with non-severe unclassified fever at the community level in the Democratic Republic of the Congo: A cluster-randomized, community-based non-inferiority trial. PLoS Med. 2018 Apr 17;15(4):e1002552. doi: 10.1371/journal.pmed.1002552. eCollection 2018 Apr. PMID 29664951
- [Derived] van Boetzelaer E, Ho LS, Gutman JR, Steinhardt LC, Wittcoff A, Barbera Y, Ngoy P, Harvey SA, Mullany LC. Universal versus conditional three-day follow up visit for children with uncomplicated fever at the community level: design of a cluster-randomized, community-based, non-inferiority trial in Tanganyika, Democratic Republic of Congo. BMC Pediatr. 2017 Jan 26;17(1):36. doi: 10.1186/s12887-017-0792-1. PMID 28122542